CLINICAL TRIAL: NCT05009875
Title: Food Trial Evaluating the Efficacy of SBD111 Versus Placebo for the Clinical Dietary Management of the Metabolic Processes of Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solarea Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SOL-SYNBIOTIC-2021
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBD111 (Experimental)
  Interventions: Other: Medical Food SBD111
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Medical Food SBD111 — Two capsules administered twice daily with morning and evening meals for 52 weeks
  Arms: SBD111
Other: Placebo — Two capsules administered twice daily with morning and evening meals for 52 weeks
  Arms: Placebo

SUMMARY:
The aim of the trial is to determine if the SYNBIOTIC (prebiotic and probiotic), provided twice daily (capsule) will help support skeletal health in otherwise healthy postmenopausal women in the early years postmenopause (1-6 years post last menstruation) over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Stated availability throughout entire study period (12 months) and willingness to fulfill all details of the protocol
* In early postmenopause (at least 1 year but a maximum of 6 years since the last menstruation)
* At least 6-months since the last intake of hormone replacement therapy
* Dual energy X-ray absorptiometry (DXA)-derived Bone Mineral Density (BMD) T-score of greater than -2.5 at the lumbar spine (L1-L4), femoral neck, and total hip but no site with BMD ≤ -2.5
* Body Mass Index between 18.5 and 35 kg/m2
* Normal levels of serum calcium (<11mg/dL)
* Normal cardiovascular parameters (systolic blood pressure ≤ 155 mm Hg, diastolic blood pressure ≤ 95 mm Hg) healthy and medication controlled

Exclusion Criteria:

The presence of any of the following criteria will exclude the participant from participating in the study:

* History of other bone disorders (eg. Paget's disease, or osteomalacia, osteogenesis imperfecta, osteopetrosis, osteoporosis, etc.)
* Women who have had cancer and were treated with radiation therapy, anti-estrogen therapy, hormonal therapy, or aromatase inhibitors
* Any history of bone or colon cancer
* Autoimmune disorders (rheumatoid arthritis, Hashimoto's disease, Graves' disease, ect), uncontrolled type 2 diabetes, gastrointestinal disorders (ulcerative colitis, Crohn's disease, inflammatory bowel disease, irritable bowel syndrome), kidney disease or dysfunction or any other medical condition that could interfere with the conduct of the study.
* History of chronic antibiotic use
* History of bariatric surgery
* History of partial colectomy
* Women with spine abnormalities that would prohibit assessment of BMD
* Women who have undergone hip joint replacement
* Women who have undergone a partial hysterectomy
* Women with untreated hyperparathyroidism
* Women previously treated with calcitonin, estrogens, estrogen derivatives, selective estrogen receptor modulators (SERMs), tibolone, progestins, anabolic steroids, or daily glucocorticoids in the past 6 months
* Women treated with bisphosphonates or strontium in the past 5 years
* Women previously treated with PTH, PTH analogs, gallium nitrate, romosozumab or denosumab
* Per-oral use of corticosteroids
* Smoking or use of nicotine products within the past 6-months
* Any disease, that by the investigator's judgement, could interfere with the intestinal barrier function
* Participation in other bone, diet, autoimmune, or gastrointestinal related clinical trials in the last 6 months
* Desire and/or plans on changing current diet and/or exercise regime during the participation of this trial
* Pregnancy or lactation
* Consumption of dietary supplements (probiotics, prebiotics) in the month prior to or during study (if participant is willing to stop taking these for 1-month, they can be enrolled after a 1-month washout period)
* Consumption of antibiotics in the past 2 months (if participant is placed on an antibiotic after enrolment in the study, will be subject to a per protocol analysis)

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Lumbar Spine Bone Mineral Density (BMD) from baseline to 52 weeks | Change in Bone Mineral Density (BMD) from baseline to 52 weeks
  Change in Bone Mineral Density (BMD) at lumbar spine following an administration period of 52 weeks and measured by DXA

SECONDARY OUTCOMES:
Change in Bone Mineral Density (BMD) at the femoral neck from baseline to 52 weeks | Change in Bone Mineral Density (BMD) from baseline to 52 weeks
  Change in Bone Mineral Density (BMD) at the femoral neck following an administration period of 52 weeks and measured by DXA
Change in Bone Mineral Density (BMD) at the hip from baseline to 52 weeks | Change in Bone Mineral Density (BMD) from baseline to 52 weeks
  Change in Bone Mineral Density (BMD) at the hip following an administration period of 52 weeks and measured by DXA
Change in volumetric BMD (vBMD) measured by quantitative computed tomography (QCT) at the lumbar spine from baseline to 52 weeks | Change in volumetric BMD (vBMD) from baseline to 52 weeks
  Change in volumetric BMD (vBMD) measured by quantitative computed tomography (QCT) at the lumbar spine (L1-L2 or L1-L4) from baseline to 52 weeks
Change in circulating C-Reactive Protein (CRP) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating C-Reactive Protein (CRP) from baseline to 52 weeks
Change in circulating Interleukin-17 (IL-17) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating Interleukin-17 (IL-17) from baseline to 52 weeks
Change in circulating Tumor Necrosis Factor (TNF) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating Tumor Necrosis Factor (TNF) from baseline to 52 weeks
Change in circulating Interleukin-4 (IL-4) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating Interleukin-4 (IL-4) from baseline to 52 weeks
Change in circulating receptor activator of nuclear factor kappa beta ligand (RANKL) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating receptor activator of nuclear factor kappa beta ligand (RANKL) from baseline to 52 weeks
Change in circulating Interferon gamma (IFNy) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating Interferon gamma (IFNy) from baseline to 52 weeks
Change in circulating C-terminal telopeptide of type 1 collagen (CTX) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating C-terminal telopeptide of type 1 collagen (CTX) from baseline to 52 weeks
Change in circulating Procollagen 1 Intact N-Terminal Propeptide (P1NP) from baseline to 52 weeks | Change from baseline to 52 weeks
  Change in circulating Procollagen 1 Intact N-Terminal Propeptide (P1NP) from baseline to 52 weeks
Safety as assessed by incidence of adverse events and serious adverse events | Change from baseline to 52 weeks
  Safety as assessed by incidence of adverse events and serious adverse events from baseline to 52 weeks
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 1-week
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 1-week
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 2-weeks
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 2-weeks
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 3-weeks
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 3-weeks
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 4-weeks
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 4-weeks
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 3-months
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 3-months
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 6-months
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 6-months
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 9-months
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 9-months
Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) | Change from baseline to 12-months
  Gastrointestinal tolerability as measured by Gastrointestinal Tolerability Questionnaire (GITQ) from baseline to 12-months
Change from baseline in the global Menopause Rating Scale (MRS) | Change from baseline to 3-months
  Change from baseline in the global Menopause Rating Scale (MRS) from baseline to 3-months
Change from baseline in the global Menopause Rating Scale (MRS) | Change from baseline to 6-months
  Change from baseline in the global Menopause Rating Scale (MRS) from baseline to 6-months
Change from baseline in the global Menopause Rating Scale (MRS) | Change from baseline to 9-months
  Change from baseline in the global Menopause Rating Scale (MRS) from baseline to 9-months
Change from baseline in the global Menopause Rating Scale (MRS) | Change from baseline to 12-months
  Change from baseline in the global Menopause Rating Scale (MRS) from baseline to 12-months

OTHER OUTCOMES:
Change in gut microbiome composition and function from baseline | Change from baseline to 6-months
  Change in gut microbiome composition and function from baseline to 6-months
Change in gut microbiome composition and function from baseline | Change from baseline to 52-weeks
  Change in gut microbiome composition and function from baseline to 12-months
Change in body composition measured by DXA | Change from baseline to 52-weeks
  Change in body composition measured by DXA from baseline to 52-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- RDC Clinical, Newstead, Queensland, Australia